CLINICAL TRIAL: NCT06279741
Title: Phase I Single Arm, Dose Escalating and Phase II Double Blind, Randomized, Placebo-controlled, Dose Finding Clinical Trial Assessing Safety and Efficacy of Intratracheal Administration of Allogeneic Umbilical Cord Mesenchymal Cells-derived Extracellular Vesicles in Preventing Bronchopulmonary Dysplasia in Extremely Preterm Newborns
Brief Title: Safety and Efficacy of MSC-EVs in the Prevention of BPD in Extremely Preterm Infants
Acronym: EVENEW
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EXO Biologics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EVENEW; 2022-500293-34 (EudraCT Number); U1111-1291-0283 (Other: Universal Trial Number)
Record Dates: First submitted 2024-02-01; First posted 2024-02-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: EXOB-001; Extracellular vesicles; Bronchopulmonary dysplasia; Extremely premature neonates; Lung inflammation
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Pneumonia | interventions — Suspensions

STUDY DESIGN:
Intervention Model Description: Phase 1 is an open-labelled, dose-escalated, and single-arm of EXOB-001. Phase 2 is a randomised, double-blind, placebo-controlled, and dose-finding of EXOB-001.
Who Masked: Participant, Investigator
Masking Description: Phase 1 is an open-label, dose-escalation and single-arm study. In phase 2, Investigators will remain blinded to each subject's assigned treatment throughout the study. The Sponsor will put in place procedures to maintain this blind. Indeed, to ensure the blinding of the groups, the preparation and administration of the test product will be organized by different teams. In the event of a Quality Assurance audit, the auditor(s) will be allowed access to unblinded study treatment records at the site(s) to verify that randomisation/dispensing has been done accurately. Blinding will be broken by the Investigator for emergency purposes only, where knowledge of the blinded treatment could influence further subject care. In addition, subjects will be unblinded for safety reports, as per regulatory requirements. Study blind will be broken after the database lock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EXOB-001 (Phase 1) (Experimental): EXOB-001 will be administered via the endotracheal route in an already intubated newborn. EXOB-001 will be administered in three dose levels (low dose, medium dose and high dose) with one or three administrations.
  Interventions: Biological: Endotracheopulmonary Instillation, Suspension
- Active group 1 EXOB-001 (Phase 2) (Experimental): In phase 2, active group 1 consists of administering the first (out of two) of the safest selected dose/regimen of EXOB-001 based on phase 1 interim results.
  Interventions: Biological: Endotracheopulmonary Instillation, Suspension
- Active group 2 EXOB-001 (Phase 2) (Experimental): In phase 2, active group 2 consists of administering the second (out of two) of the safest selected dose/regimen of EXOB-001 based on phase 1 interim results.
  Interventions: Biological: Endotracheopulmonary Instillation, Suspension
- Placebo (Phase 2) (Placebo Comparator): In phase 2, the saline solution for infusion is used as a placebo.
  Interventions: Biological: Endotracheopulmonary Instillation, Suspension

INTERVENTIONS:
Biological: Endotracheopulmonary Instillation, Suspension — The endotracheal administration can be either by endotracheal tube instillation using a 5 French end-hole catheter or by endotracheal tube instillation using the secondary lumen of a dual lumen endotracheal tube.
  The dose is adjusted to body weight and the endotracheal administration will be performed in an already intubated newborn infant.
  Other Names: Endotracheopulmonary instillation

SUMMARY:
The phase 1/2 trial aims to evaluate the safety and efficacy of EXOB-001 consisting of extracellular vesicles derived from umbilical cord mesenchymal stromal cells in the prevention of bronchopulmonary dysplasia (BPD) in extremely premature neonates. The study population includes babies born between 23 and 28 (27 + 6 days) weeks of gestational age and body weight between 500g and 1,500 g. Thirty-six subjects will receive one or three administrations of the three doses of EXOB-001 via the endotracheal route in phase 1. In phase 2, two dosages based on the results of phase 1 will be selected and a total of 203 subjects will be randomised to receive either EXOB-001 or placebo (saline solution).

Infants will be followed up to 2 years of corrected age (end of study).

DETAILED DESCRIPTION:
Bronchopulmonary Dysplasia (BPD) is a chronic severe multifactorial respiratory disease that affects extremely premature infants and is the most common and severe consequence of preterm birth. BPD is associated with disrupted alveolarization and microvascular development, resulting in abnormal gas exchange and lung mechanics. BPD has a multifactorial aetiology, with pre-, peri-, and postnatal mechanisms causing inflammation and injury and resulting in the disruption of the lung's development with the insurgence of an aberrant repair mechanism.

EXOB-001 consists of a population of EVs smaller than 0.22 μm in diameter, containing proteins and nucleic acids, enclosed in a double layer of phospholipids with integral and surface-bound proteins as the main components. EVs exert anti-inflammatory and immunomodulatory activity by reducing the release of proinflammatory cytokines and reducing the recruitment of immune cells in the lung. Current evidence shows that EVs can modulate macrophage phenotype, and this is relevant for BPD, because of the role macrophages have in its pathogenesis.

Two hundred sixty-five (265), 40 in phase 1 (to reach 36 evaluable subjects) + 225 in phase 2 (to reach 203 evaluable subjects), extremely preterm infants at risk of developing BPD with 23 weeks up to 28 (27 weeks+6 days) weeks of gestational age and birth weight between 500g and 1,500g and being endotracheally intubated between postnatal day 3 and day 10 receiving mechanical ventilation with FiO2 > 25%.

Phase 1 will start with cohorts with a single administration starting with a low dose up to a high dose and thereafter start the escalation of cohorts with 3 administrations starting with a low dose up to a high dose. In the case of 3 endotracheal administrations, there will be a window of 24 hours between the administrations (the maximal duration of the treatment with EXOB-001 will be 48 hours).

Phase 2 includes 2 groups with selected dosage levels and regimen of EXOB-001 based on phase 1 interim results. Subjects will be randomised (2:2:1) to receive either EXOB-001 or placebo (saline solution).

ELIGIBILITY:
Inclusion Criteria:

* From birth up to 10 days chronological age.
* From 23 weeks up to 28 weeks (27 week+6 days) gestational age at birth.
* Birth weight ≥ 500g but ≤1500g.
* Endotracheally intubated and receiving mechanical ventilation with FiO2 > 25% anytime between 3 and 10 days postnatally or needing re-intubation due to respiratory complications, - Not expected to be extubated within the next 24/48 hours after enrolment.
* Written informed consent from parents/legally designated representative.

Exclusion Criteria:

* Surfactant administration less than 24 hours prior to (first) IMP administration.
* Has a congenital heart defect, except for patent ductus arteriosus (PDA), atrial septal defect or a small/moderate, restrictive ventricular septal defect.
* Has a serious malformation of the lung, such as pulmonary hypoplasia/aplasia, congenital diaphragmatic hernia, or any other congenital lung anomaly.
* Being treated with inhaled nitric oxide.
* Has a known chromosomal abnormality (e.g., Trisomy 18, Trisomy 13, or Trisomy 21) or a severe congenital malformation (e.g., hydrocephalus and encephalocele, trachea-oesophageal fistula, abdominal wall defects, and major renal anomalies).
* Has had a known severe congenital infectious disease (i.e., herpes, toxoplasmosis rubella, syphilis, human immunodeficiency virus, cytomegalovirus, etc.).
* Active systemic infection, severe sepsis, or septic shock at Screening up to baseline (phase I) or randomization (phase II).
* Underwent a surgical procedure (requiring admission to an operating room) within 72 hours before baseline (phase I)/randomization (phase II) or who is anticipated to have a surgical procedure (requiring admission to an operating room) within 72 hours before or following baseline (phase I)/randomization (phase II).
* Has had a Grade 3 or 4 intraventricular haemorrhage (IVH).
* Has active pulmonary haemorrhage.
* Has periventricular leukomalacia (PVL).
* The subject is currently participating in any other interventional clinical study.
* The subject is, in the opinion of the Investigator, so ill that death is inevitable, or is considered inappropriate for the study such as an infant that received thoracic compressions and/or adrenaline administration during stabilization in the delivery room and for any reason(s) other than those listed above.

Max Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 265 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (phase 1) | From EXOB-001 administration up to 36 weeks post-menstrual age (PMA)
  The proportion of subjects exhibiting acute and short-term safety of the intratracheal administration of EXOB-001 (single dose or multiple doses at different dose levels).
Number of subjects with BPD grade II-III incidence rate per groups (phase 2). | 36 weeks PMA
  BPD grade II-III incidence rate per group assessed at 36 weeks PMA. The severity of BPD is assessed according to the modified NICHD severity grading (Grade I to IIIA) definition.

SECONDARY OUTCOMES:
Assessment of medium-term safety of EXOB-001 (phase 1/2) | From EXOB-001 administration to hospital discharge (between 36 and 40 weeks PMA)
  The proportion of subjects experiencing treatment-emergent adverse events (TEAE) from EXOB-001 administration up to hospital discharge
Number of subjects with dose-limiting toxicity (DLT) (phase 1) | 6 hours and 24 hours after EXOB-001 administration
  DLT is measured as:
  * cardiorespiratory decompensation;
  * decrease in SpO2/FiO2 ratio;
  * stable increase in required mean airway pressure >3 cm H2O;
  * death,
  * anaphylactic reaction.
  * any serious adverse reaction (SAR) considered as at least possibly related to EXOB-001 administration.
Number of subjects needing for oxygen and ventilation for BPD incidence (phase 1/2) | 28 days chronological age, 36 weeks PMA, 40 weeks PMA
  The number of subjects needing oxygen and ventilation support.
Assessment of immune markers (phase 2) | Baseline (before EXOB-001 administration), baseline + 24 hours before EXOB-001 administration, baseline + 72 hours if the the subject is still intubated
  To test immune markers in the tracheal aspirate fluid.
Assessment of BPD incidence and severity (phase 1/2) | 28 days of chronological age, 36 weeks PMA and 40 weeks PMA
  The number of cases and severity of BPD were measured according to different definitions (modified NICHD severity grading (Grade I to IIIA), Jobe and Bancalari 2001, and Isayama 2017).
Safety evaluation (phase 1/2) | From enrolment to 2 years of corrected age (end of study)
  All adverse events (AEs) and serious adverse events (SAEs) (including case fatalities), both related and non-related.
Assessment of lung ultrasound score (phase 1/2) | From baseline to 2 years of corrected age (end of study)
  The lung ultrasound score (LUS) aims to assess lung development in all groups by lung ultrasound at different time points.
  Each lung is divided into 3 areas (upper anterior, lower anterior, lateral), and each area will be evaluated by assigning a value ranging from 0 to 3 to each zone, with a consequent overall value ranging between 0 and 18 in all infants scanned on the anterior and later thorax, and also another score (called extended lung ultrasound score or eLUS) in those infants scanned posteriorly ranging between 0 and 30.
  The lung ultrasound scores were assigned as follows:
  * 0, indicates an A-pattern (defined by the presence of the only A-lines);
  * 1, indicates a B-pattern (defined as the presence of ≥3 well-spaced B-lines);
  * 2, indicates severe B pattern (defined as the presence of crowded and coalescent B lines with or without consolidations limited to the subpleural space);
  * 3, indicates extended consolidations.
Number of subjects with complications of prematurity (phase 1/2) | From baseline to 2 years of corrected age (end of study)
  To assess all known complications of prematurity, concomitant treatments/procedures/therapies in all groups.
Assessment of the respiratory morbidity (phase 1/2) | From hospital discharge to 2 years of corrected age (end of study)
  To evaluate the respiratory morbidity by the Liverpool Respiratory Symptom Questionnaire in all groups at different time points.
  Parents are asked to consider respiratory symptoms over the last 3 months, with questions being scored on a five-point Likert scale from ''not at all'' (score 0) to ''every day'' (score 4). A score for each domain and the complete questionnaire is calculated.
Assessment of neurodevelopment (phase 1/2) | From hospital discharge to 2 years of corrected age (end of study)
  To evaluate the neurodevelopmental condition by the ASQ3 questionnaire in all groups with age-specific questionnaires at different time points. The neurodevelopment will be assessed by five domains: communication, gross motor, fine motor, problem-solving, and personal-social.
  Parents will fill out each item and indicate whether the baby is doing the activity regularly (10 points), sometimes (5 points), or not yet (0 points).
  The total score of each developmental area is compared to the area cut-offs.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice De Vos, M.D., Ph.D., Study Chair — EXO Biologics SA
Locations (8):
- Belgium (3):
  - Cliniques Universitaires Saint-Luc (UCLouvain), Brussels
  - ISPPC CHU Charleroi, Charleroi
  - Clinique CHC Montlégia, Liège
- Italy (5):
  - AOU Careggi, Florence
  - IRCCS Instituto Giannina Gaslini, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - AOU Policlinico di Modena, Modena
  - Unità di Fase I della UOC Terapia Intensiva e Patologia Neonatale, Assistenza Neonatale (TINI) dell'Azienda Ospedale Università di Padova, Padua